CLINICAL TRIAL: NCT07121166
Title: Effectiveness of a Tele-group Cognitive Behavioural Family Intervention (tgCBFI) for People With Schizophrenia and Their Families: a Mixed-method Study
Brief Title: Tele-group Cognitive Behavioural Family Intervention for Individuals With Schizophrenia and Their Families
Acronym: tgCBFI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: health bureau, hong kong (Unknown)
Responsible Party: Principal Investigator, Dennis Chak Fai Ma, Assistant Professor of Practice, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20241014006
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia and Related Disorders
Keywords: CBT; family intervention; schizophrenia; telehealth
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tgCBFI group (Experimental): Participants in this group will receive a six-week online group intervention programme and integrated community psychiatric care with psychiatric outpatient follow-up.
  Interventions: Behavioral: tgCBFI programme
- Treatment as Usual (TAU) group (Active Comparator): Participants in this group will receive integrated community psychiatric care with psychiatric outpatient follow-up
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: tgCBFI programme — a six-week online group intervention programme for dyads of service users and caregivers
  Arms: tgCBFI group
Behavioral: Treatment as Usual (TAU) — Integrated community psychiatric care with psychiatric outpatient follow-up
  Arms: Treatment as Usual (TAU) group

SUMMARY:
This mixed-method study comprises a RCT with a twelve-week post-intervention follow-up and focus group interviews. The RCT study aims to examine the effectiveness of delivering the tgCBFI programme to dyads of people with schizophrenia and their family caregivers, while the focus group interviews aim to qualitatively study the benefits of the tgCBFI programme from the service users and their family caregivers to provide a more in-depth understanding and complement the quantitative data. The main questions it aims to answer are: Does this online tgCBFI programme reduce the expressed emotion experienced and positive and negative symptoms of individuals with schizophrenia? Does this online tgCBFI programme reduce the perceived care burden and level of mood disturbances of family caregivers?

DETAILED DESCRIPTION:
Recent network meta-analyses revealed that family interventions were superior to other psychosocial interventions in relapse prevention of people with schizophrenia. The current approaches to family intervention for schizophrenia are to provide support and offer psychoeducation and skill training for family caregivers, such as family psychoeducation and mutual support groups, and work with the whole family, stressing family structure, interaction, and dynamics, such as systemic therapy. A previous meta-analysis revealed that familial expressed emotion (EE), particularly critical comments, is a robust predictor of schizophrenic relapse, and it is one of the therapeutic foci of the family intervention to benefit the recovery of service users with schizophrenia. A proposed cognitive model of caregiving suggested that cognitive reappraisal, including reattribution of self-control on caregiving and reattribution of service users' control on illness progression, is one of the recommended therapeutic components to assist family caregivers in relieving their mood disturbances as well as negative expressed emotion. A framework of cognitive behavioural therapy (CBT) for service users with psychosis and their family caregivers has also been suggested to improve the clinical outcomes of the service users and extend the individual CBT to the family group. Built upon these two mainstream approaches of behavioural and structural family interventions, cognitive behavioural family intervention (CBFI) focuses on cognitive appraisals in family relationships between service users and their families, aligning with the proposed cognitive model of caregiving in resolving the two negative attrition-emotion pathways. A previous meta-analysis indicates that CBFI is superior to treatment as usual (TAU) in reducing the severity of positive and negative symptoms of people with schizophrenia immediately following the intervention. Recent systematic reviews supported that telepsychiatry/telehealth is a feasible and acceptable approach for people with severe mental illness and their family caregivers. This tgCBFI programme is a brief, novel group CBT-based family intervention using a telehealth delivery mode (i.e., via Zoom) to care for people with schizophrenia and their family caregivers in the community.

ELIGIBILITY:
I. Individuals with schizophrenia-spectrum disorders

Inclusion Criteria:

* current diagnosis of schizophrenia-spectrum disorders, based on ICD-10 made by the treating clinicians,
* aged 18-64, and
* able to read and write Chinese

Exclusion Criteria:

* having co-morbidity of learning disability, organic/neurological conditions, or substance use disorder, and
* living in a hostel

II. Family caregivers

Inclusion Criteria:

* aged 18 or above,
* able to read and write Chinese,
* live with service users, and
* nominated by the service users

Exclusion Criteria:

* having active psychiatric conditions

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Expressed emotion experienced by the service users as assessed by the Concise Chinese Level of Expressed Emotion Scale (CCLEES) | From enrollment to twelve-week post-intervention follow-up
  It has twelve items using a four-point Likert scale with three subscales. The total score ranges from 12 to 48, and a higher score indicates a higher level of familial expressed emotion.

SECONDARY OUTCOMES:
Positive and negative symptoms of service users as assessed by the Positive and Negative Syndrome Scale (PANSS) | From enrollment to twelve-week post-intervention follow-up
  It has thirty items using a seven-point Likert scale with three subscales. The subscale scores of positive and negative symptoms range from 7 to 49, while that of general psychopathology ranges from 16 to 112. A higher score indicates a higher level of severity of psychiatric symptoms.
Perceived care burden of family caregivers as assessed by the Family Burden Interview Schedule (FBIS) | From enrollment to twelve-week post-intervention follow-up
  It has 25 items using a three-point Likert scale with six subscales. The total score ranges from 0 to 50. A higher score indicates a higher level of perceived family care burden.
Mood disturbances of family caregivers as assessed by the Hospital Anxiety and Depression Scale (HADS) | From enrollment to twelve-week post-intervention follow-up
  It comprises fourteen items using a four-point Likert scale with two subscales. The subscale scores of depression and anxiety range from 0 to 21. A higher score indicates a higher level of mood disturbance.
Service satisfaction of participants from the tgCBFI group as assessed by the Client Satisfaction Questionnaire (CSQ-8) | within one week after the intervention
  It consists of eight items using a four-point Likert scale. The total score ranges from 8 to 32. A higher score indicates a higher level of service satisfaction.
Qualitative feedback from the participants in the tgCBFI group as assessed by focus group interviews | within one month after the intervention
  For each interview, a group of eight participants will be interviewed for up to 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chak Fai Ma, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon reasonable request to the corresponding author after the study articles are published.